# National Taipei University of Nursing and Health Sciences Doctoral Dissertation Proposal

## **School of Nursing**

The Effect of a Yoga Intervention for Reducing Stress among People Living
with HIV in Indonesia: A Randomized Controlled Trial
(Study Protocol and Statistical Analysis Plan)

Jufri Hidayat

Advisor: Miao-Yen Chen RN, PhD

NCT Number: NCT05503680

Document date: January 7th, 20223

## 1. Yoga protocol intervention

Participants in the yoga group engaged in eight biweekly online Hatha yoga classes for 120 minutes each at home. Classes began with 15 minutes of sitting meditation; breathing exercises; shoulder, neck, and back stretches; and sun salutations (either seated or standing). Following that, ten minutes of standing poses, fifteen minutes of balancing poses, and ten minutes of abdominal and back-bend positions will be performed. After 10 minutes of cool-down stretches and a final time of rest, all sessions was concluded. Physical postures and supportive props were modified to accommodate participants of all abilities. Participants was given an honorarium of Rp 50.000 or 3.49 USD at the baseline and final assessments. The full version of the yoga protocol is available in appendix III.

Table 3: Yoga protocol

| Position | Main content | Length time |
|-------------------|------------------------------------------|-------------|
| 1. Warm-up | (1) Seated meditation, (2) Alternate (3) | 10 minutes |
| | Nostril breathing, (4) Bellows breath, | |
| | (5) Shoulder/neck stretches, (6) Cat-cow | |
| | forward fold, (7) Sun salutations. | |
| 2. Standing poses | (1) Warrior one, (2) Warrior two, (3) | 10 minutes |
| | Triangle, (4) Extended side angle, (5) | |
| | Reverse warrior, (6) High lunge with | |
| | twist. | |
| 3. Balance poses | (1) Tree pose, (2) Standing holding | 10 minutes |
| | knee, (3) Modified warrior three (chair | |
| | support), (4) Half-moon. | |

| 4. | Abdominal and back | (1) Bird-dog, (2) Side plank, (3) Bridge, | 10 minutes |
|---|---|---|---|
| | bends | (4) Cobra, (5) Sphinx, (6) Baby position | |
| 5. | Meditation | Full lotus, half lotus, Burmese | 10 minutes |
| 6. | Cool down | (1) Twist, (2) Cobbler's pose, (2) Hip (3) Stretches, (4) Corpse pose, (5) Side- | 10 minutes |
| | | lying, (6) Seated on. | |

# The Yoga Protocol



A Hatha Yoga protocol to reduce stress among people living with HIV

Jufri Hidayat Doctoral student



National Taipei University of Nursing and Health Sciences

| Yoga intervention for stress reduction among people living with HIV |
|---|
| Estimated length of time per session: 60 minutes |
| Created by: |
| Jufri Hidayat |
| Doctoral student at National Taipei University of Nursing and Health Sciences |
| Supervisor: |
| Miao-yen Chen |
| Associate Professor at National Taipei University of Nursing and Health Sciences |

All rights reserved

**Preface** 

This 60-minute yoga protocol was developed for participants in the research project, "The

effect of a yoga intervention for reducing stress among people living with HIV during the covid-

19 pandemic in Indonesia, a randomized controlled trial."

You have been given a copy of this protocol because you are an HIV positive person and are

undertaking a yoga intervention program to reduce stress. This protocol has an instructor and

pictures of yoga poses to help you to practice yoga correctly. Share this protocol with your

family, friends, or community who might need help to recover from stress related to HIV.

Jufri Hidayat

**Doctoral student** 

February 3<sup>rd</sup>, 202

| Position | Activity/purpose | Action plan | | |
|---|---|---|---|---|
| Warm up (15 minutes) | Activity: (1) Seated meditation, (2) Alternate | | | |
| | nostril breathing, (3) Bellows breath, (4) Shoulder/neck stretching, (5) Cat-cow forward fold, (6) Sun-salutation. | 200 0000 | 2000 0000 | 200 |
| | Maximum duration: 15 minutes Purpose: | | | The state of the s |
| | Warming up for hatha yoga aims to | | | <u> </u> |
| | help participants to prepare their | 1. Seated meditation | 2. Alternate nostril | 3. Bellows breath |
| | minds to be centered, calm, and focused. | Sit on yoga mat with | breathing Sit on yoga mat with legs | Instruction: |
| | A distracted mind prevents | legs crossed and body | crossed and body | Sit as in seated meditation, |
| | participants from reaping the deepest | relaxed. | relaxed. Place left hand | with shoulders relaxed. |
| | psychological and spiritual benefits | Place both hands on | on left knee. Raise your | Take a few deep breaths, |
| | from yoga practice. | legs. Keep your lower | right hand towards your | breathing in and out from |
| | | jaw parallel to the | nose and exhale | nose. With each inhale, |
| | Equipment: | ground. Relax your | completely. Use your | expand your belly fully |
| | Yoga mattress, chair, sport clothes, chair | abdomen, feet, pelvis, | right thumb to close your | with your breath. Begin |
| | | and shoulders. Sit | right nostril while you | bellows breath by exhaling |
| | | upright so your spine is | inhale through the left | forcefully through your nose at the rate of one |
| | | centered between your left and right shoulders, | nostril. Then close your left nostril with your | breath per second. These |
| | | with your eyes closed. | index finger as you open | are a series of short sharp |
| | | Observe the breath | the right nostril, exhaling | exhales, with passive |

through the right side. inhalation happening in coming in and going out, letting thoughts Next inhale through your between. Make sure the float away like logs right nostril, then close it breath comes from your rolling down the river. as you open the left diaphragm, with your belly nostril and exhale moving in and out. head, through the left side. This neck, shoulders, and chest is one cycle. Repeat 5 times. 5. Cat-cow forward fold 4. Shoulder/neck 6. Sun salutation stretching Instruction: Instruction: Begin on Instruction: sit as in seated meditation. Place your hands and knees in Begin in a standing one of your hands the table pose, with your position with your feet behind your back with spine relaxed. As you slightly apart and parallel the other hand on top of exhale, come into cat to each other, your palms turned out, and shoulders your head. With the pose by rounding your hand on your head, spine outward like a cat relaxed. Then follow this gently pull your ear arching its back, tucking sequence of positions: toward your shoulder. your tailbone in, and mountain pose (i.e., Feel the stretch at the drawing your stomach in. standing with the palms of side of the neck. Hold it Next, as you inhale, your hands facing towards for 20 seconds and your body alongside your move into cow pose by repeat three times. Then lifting your sit bones thighs), Inhaling, lift both

| repeat these steps for | upward, pressing your | arms up. Exhaling, fold |
|---|---|---|
| the other side. | chest down and forward, | forward at the hips |
| the other side. | lifting your head up and | bringing your hands down |
| | allowing your belly to | to the mat. Step the right |
| | sink. | leg back and lunge. Then |
| | Relax your shoulders | step the left leg back in |
| | away from your ears, | plank, keeping body |
| | gazing straight ahead. | parallel to the floor. Then, |
| | gazing straight anead. | |
| | | bending yourelbows bring the chest down to the |
| | | l l |
| | | ground. Push up with your |
| | | hands, straightening the |
| | | elbows and sliding |
| | | forward into up dog. Curl |
| | | the toes under, press down |
| | | on feet and hands, lifting |
| | | your hips up. Straighten |
| | | elbows and knees. Then |
| | | step your right foot |
| | | forward so your right foot |
| | | is parallel with your hands. |
| | | Bring left foot up to the |
| | | right foot andyou are |
| | | standing flexed at the hips |
| | | in forward fold. Inhaling |
| | | and standing up, swoop |
| | | the arms out to the sides |
| | | and above your head. |
| | | Bring the palms together |

| | | | | and lower them to your heart in namaste and back to mountain pose. The yoga instructor will demonstrate how to do this. |
|---|---|---|---|---|
| Standing | Activity: | | | |
| pose | (1) Warrior one, (2) Warrior two, (3) | | | |
| (10 minutes) | Triangle, (4) Extended side angle, (5) Reverse warrior, (6) High lunge with twist. Maximum duration: 10minutes | 6000 G6600 | 00000 0000 | 2000<br>2000<br>2000 |
| | Purpose: | | | |
| | Strengthen and stretch all muscle | 1. Warrior one | 2. Warrior two | 3. Triangle |
| | groups in the legs, particularly the | Instruction: | Instruction: | Instruction: |
| | thighs, hamstrings, buttocks, calves | Begin by standing. Then | Start in standing (i.e., | Begin standing, then |
| | and ankles. | extend your right foot | mountain) pose. Step | spread your feet apart to |
| | Build balance and stability and Supply the stability and | forward. Bend your right knee into a lunge | your right foot out to your side with your feet | a position wider than your shoulders. Bend |
| | improve flexibility. | with your feet parallel | wider than shoulder | your left leg slightly and |
| | • Reduce stress and promote better sleep. | and toes pointing | length apart in a five- | raise your arms out from |
| | sicep. | forward. Keep your left | pointed star position. | your sides until they are |
| | | leg straight behind you | Turn your right foot out | parallel to the ground, |
| | | and turn your left heel | to the right at a 45 degree | forming a "T" shape. |
| | | approximately 45 | angle. Bend your right | Place your left hand |

| degrees outward. Raise your arms straight above your head, keeping shoulders down. Squeeze your shoulder blades together and pull them downward. Lift your chin to gaze at your hands overhead. Hold this pose, then lower your arms and repeat on the left side. | knee until the knee is above your ankle. Extend your arms parallel to the ground. Relax your shoulders downwards. Turn your left foot out 90 degrees, then bend your right knee into a lunge. Be sure to keep the knee of your right leg above your ankle and pointing past your toes. Turn your head to the left and look beyond your fingers. Repeat this on the other side. | either on your left leg or touching the mat in the front of your left foot. Raise your right arm, extending it overhead and hold. Then repeat on the other side. |
|---|---|---|
|---|---|---|



| hand down to the floor<br>or to a yoga block<br>placed in front of your<br>foot. |
|---|

## Balance pose

## Activity:

(1) Tree pose, (2) Standing holding knee,(3) Modified warrior three (chair support), (4) Half moon.

Maximum duration: 15 minutes

#### Purpose:

- Strengthening and lengthening the muscles.
- Exploring your center of gravity and improving the body's equilibrium.
- Improving focus, concentration, and memory and relieving stress



1. Tree poses



2. Standing holding knee



3. Modified warrior 3 (Chair support)

#### Instruction:

Begin in mountain pose. Shift your weight onto your left leg. Bend your right knee and place your right foot on the inside of your left leg, either above or below the knee joint, pressing your foot against your inner thigh. Pull your left hip in over your left foot (use chair or wall to help balance if needed). Lengthen your spine, loosen shoulders and tuck your chin slightly in and back, bringing

## Instruction:

Begin in mountain pose. Place your left hand on your hip. Moving very slowly, draw your right knee up towards your chest. With your right hand, hug your knee to your chest. Lengthen your spine, tightening the muscles of your left side and abdomen. Stiffen your left leg, but do not lock your knee. Drop your right hip slightly until it is in line

#### Instruction:

Begin with warrior one on the right side. Bring your palms together and begin to lean forward. Lift the left leg off the floor, keeping the body, arms, and raised left leg parallel to the floor, flexing the toes. Strenghten the standing leg and your arms. Fix your gaze looking down, hold the pose and breathe. Then lower your leg back down into warrior 1 position. then practice on the other side.

| your hands in front of your heart (prayer position). Stay in this pose for 30 seconds or 1 minute, then repeat on the other side. | with your left hip. Hold for 1 minute. |
|---|---|
| 4. Half-moon pose (chair support) Instruction: Start in warrior 2 with a chair beside you. Bring your right hand to your hip and turn your head to look at the floor. Bend your front leg and shift your weight onto your front foot. Move your hand a little forward and place your forearm on the chair | |

| shoulder. Press down through your fingers to steady yourself. Lift your back leg until your thigh is parallel to the floor. Slowly turn your chest to face the right. Extend your other arm toward the ceiling. Either keep your gaze on the floor or slowly bring it to your hand above. |
|---|

| Abdominal |
|-----------|
| and back |
| bends |

## Activity:

- (1) Bird-dog, (2) Side plank, (3) Bridge, (4) Cobra, (5) Sphinx.
- (1) Coora, (3) Spinis

Duration: 10 minutes

## Purpose:

- Lengthen and strengthen spine, promoting flexibility, mobility, and good posture.
- Stretch shoulders, chest, and abdomen.
- Reduce stress and anxiety.



1. Bird-dog





Instruction: Begin with plank pose (with your weight on both forearms) and press your palms into the mat as you lift up through your shoulder). Turn onto the outside of your right foot, stacking your left foot on top of it. Rotate your entire body to face forward with your flank toward the floor. Press your right hand down, keeping your body even from heel to fingers, as you raise your left arm up toward the sky. Take 5 to 10 deep breaths.



3. Bridge

Instruction: Lying on your back, place your feet flat on the floor, with your arms next to your ribcage. Inhale and press the back of your shoulders and your feet into the floor and lift your hips. Actively press the inside of feet down and keep your knees from spreading out wide. You're your belly in and slide your shoulder blades down your back, keeping your neck neutral. You can clasp your hands

## Instruction:

Begin with hands and knees on the floor in the tabletop position, with knees under hips and hands under your shoulders. Maintain a neutral spine by firming up your abdominal muscles. Draw your shoulder blades together, raising right arm and left leg. Keeping shoulders and hips parallel to the floor, extend the back of your neck and tuck your chin into your chest to gaze down at the floor. Hold this position for a

| few seconds, then do the other side. | | behind your back. Stay in this position for 5 to 15 breaths. |
|---|---|---|
| 4. Cobra | 5. Sphinx | 6. Baby position |
| Introduction: | Introduction: Lying down | Introduction: Place |
| Lie on your stomach, | on your belly with your | your hands and knees |
| with your toes pointing | shoulders over your | on the mat. Spread your |
| straight back. Position | elbows, with your | knees the same width as |
| your hands underneath | forearms flat on the floor. | the mat and extend your |
| your shoulders, with | Bring your shoulder | big toe with your big |
| elbows close to your | blades together sliding | toe on the floor. Place |
| body. With legs engaged, | down your back and feel | your stomach between |
| pull the belly in and up, | your chest pushing | your thighs and your |
| lifting your chest from | slightly foreward. | forehead on the floor. |
| the back of your heart. | Breathe into your lower | Relax your shoulders, |
| Sticking your chest out, | back and abdomen. To | chin and eyes. If you're |
| pull your shoulder blades | come out of the pose, | not good at putting your |
| together and down along | lower your torso, | forehead on the floor, |
| the spine. Come down | bringing your elbows | put your forehead on a |
| | toward your sides and | |

| | | gradually as you exhale. Repeat that two times. | rest your forehead on your hands. | stack of fist blocks or two |
|---|---|---|---|---|
| Cool down | Activity: (1) Twist, (2) Cobbler's pose, (3) Hip stretches, (4) Corpse pose, (5) Sidelying, (6) Seated on. Duration: 10 minutes Purpose: • Gradually slow down allowing heart rate to return to normal, preventing muscle soreness. • Reduce stress and improve relaxation. | 1. Twist Instruction: Begin in seated meditation pose with right leg crossed on top of your left. Inhale and bring you right hand straight up beside your right ear. Exhale and twist your torso to the left, bringing your right elbow to the outside of your left knee and place your left palm on the floor slightly behind | 2. Cobbler's pose Instruction: Bend your knees and bring the soles of your feet together. As you let your knees fall down to either side, draw your feet in towards your body as far as you comfortably can. Press the outer edges of your feet together firmly. You can use your hands to pull | 3. Hip stretches Instruction: Lie on your back with your knees bent and feet flat on the floor. Bend your right knee until your lower leg is perpendicular to the floor. Then bring your left knee up, rotating your left leg outward at the hip so you can rest your left ankle on your right thigh just above the knee. Bring your right hand to the outside of the right thigh and pass your left |

| your sit bones. Direct<br>your gaze over your left<br>shoulder without<br>straining your neck. On<br>each inhale, lengthen<br>your spine upwards. On<br>each exhale, deepen the<br>twist slightly. | your feet together and toward your body. | hand through the opening formed by your crossed left leg. As you pull your right thigh toward your chest with your hands, press your left thigh with your left elbow. Hold for 30 seconds. |
|---|---|---|
| 4. Corpse pose | 5. Side-lying | 6. Seated on |
| Introduction: Lie on your back. Separate your legs slightly and allow your feet to fall open to either side. Bring your arms down alongside your body, at a small distance from your torso. Turn your palms to face upwards but let the fingers curl in. Tuck your shoulder blades into | Instruction: Rest on the mat on your most comfortable side. Use your arm or a folded blanket to support your head and another to separate your knees. Roll the top hip slightly forward and shift the bottom hip slightly | Instruction: This seated meditation pose is the last pose of the yoga series, exactly the same as the first one. Hold this position for one minute. |

| your back. Once you have put your limbs in | back so the hip joints are not stacked on top |
|---|---|
| place, relax completely without making an effort to holding them in | of each other. Relax<br>the belly and breathe<br>slowly and deeply. |
| position. Relax your entire body, including | Feel the breath in your body as you |
| your face. Feel the weight of your body | gently observe each inhale and exhale. |
| against the floor. | |

## 3. Statistical analysis plan

Before performing statistical procedures, all data was entered into a computer and checked for errors. To analyze the data, the researcher then used SPSS computer software version 20. The data for all variables was manually coded before using the SPSS application, including demographic characteristics of patients, the perceived stress scale results brief health status survey, and coping self-efficacy. The alpha value was set at  $\alpha$ =0.05 to determine the statistical significance of the variables. For demographic characteristics, the data analysis was descriptive statistics to identify the frequencies and percentages for categorical variables and the means and standard deviations for continuous variables. Before the statistical data processing begins, the data for independent and dependent variables was tested to determine its distribution and normality using plot histograms, logs and square roots, and checking residuals.

This study took repeated assessments over time and used a Generalized Estimating Equation (GEE) approach to model each study outcome and to predict the relationship of the variables while accounting for correlated data within the repeated measures (Hardin & Hilbe, 2007). The GEE technique, introduced by Liang and Zeger (1986), was the most often used strategy in marginal models, and it was a variation of Generalized Linear Modelling (GLM). GEE can handle correlated data with discrete, continuous, or binary outcomes. GEE is a non-likelihood or quasi-likelihood data modeling approach that specifies one of many working correlation matrix architectures to account for within-subject correlations (Liang & Zeger, 1986).